CLINICAL TRIAL: NCT06172907
Title: A Dyadic Intervention for Young Adult Patients With Cancer and Their Partner Caregivers
Acronym: YAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jamie Jacobs, Assistant Professor, Harvard Medical School Department of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-472
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Survivorship; Caregiver Burden; Psychological Distress; Coping Skills; Couples
Keywords: Young Adult Cancer; Cancer Caregiving
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Single-Arm Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young Adults Coping with Cancer Together Intervention (Other): Young adults with cancer and their partner-caregivers will attend dyadic virtual psychotherapy sessions lasting 45-60 minutes on a weekly basis for eight weeks.
  Interventions: Behavioral: Young Adults Coping with Cancer Together Intervention

INTERVENTIONS:
Behavioral: Young Adults Coping with Cancer Together Intervention — This intervention is based on cognitive-behavioral therapy and couples' therapy. It aims to improve cancer and caregiving-related self-efficacy and coping, as well as promote relationship maintenance in context of cancer. The intervention will be delivered by a trained mental health practitioner and include didactics, experiential exercises, and home practice.
  Other Names: YAD Intervention

SUMMARY:
The purpose of this pilot study is to examine the feasibility and acceptability of a brief psychotherapy intervention to improve psychosocial coping and maintain couple relationships among young adults (aged 25-39) with cancer and their caregiving partners.

DETAILED DESCRIPTION:
Young adults (YA) with cancer have unique challenges in coping, and their primary partners may experience burden and low self-efficacy related to caregiving. In this single-arm pilot trial, the investigators shall deliver an eight-session intervention to YAs with cancer and their self-identified partners who provide caregiving. The intervention is founded on principles from cognitive-behavioral therapy and couples-focused interventions, tailored for YA. The aim of the study is to assess the feasibility and acceptability of the intervention, which will inform refinements prior to a larger-scale clinical trial. This study will include 10 YAs and their partner-caregivers (N=20). Participants will complete surveys at baseline and after the intervention, and will be invited to complete optional semi-structured exit interviews.

ELIGIBILITY:
Inclusion Criteria:

* Either: (1) Currently receiving active cancer treatment (n=5) or are within two years of completing active treatment (n=5) at Massachusetts General Cancer Center (MGHCC), located in Boston, Massachusetts, United States, OR (2) are the partner of an individual between the ages of 25-39 who is currently receiving treatment at MGHCC (n=5) or who has completed cancer treatment at MGHCC within the past two years (n=5)
* Either: (1) Indicates a score ≥4 on the National Comprehensive Cancer Network (NCCN) adapted distress thermometer study screening questions, OR (2) are the partner of a participant indicating a score ≥4 on the NCCN adapted distress thermometer study screening questions
* English-speaking

Exclusion Criteria:

• Uncontrolled psychosis, active suicidal ideation, or cognitive impairment

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | 14 +/- 2 Weeks
  Feasibility will be measured by measured by participant rates of enrollment (≥50% of those eligible), participant retention (≥70% of those enrolled), and intervention attendance (≥70% attending at least 6 of 8 sessions).
Acceptability of Intervention | 14 +/- 2 Weeks
  Acceptability with be measured by satisfaction with the intervention as rated on the Client Satisfaction Questionnaire. The intervention will be deemed acceptable if ≥75% of participants report average satisfaction that exceeds the CSQ's midpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Jacobs, Ph.D., Principal Investigator — Massachusetts General Hospital; Giselle K Perez, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Emerson Hospital/MGH Cancer Center, Concord, Massachusetts
  - Mass General at North Shore Cancer Center, Danvers, Massachusetts
  - Mass General at Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: jjacobs@mgh.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team
URL: https://www.massgeneralbrigham.org/en/research-and-innovation/innovation